CLINICAL TRIAL: NCT02344056
Title: Cognition Intervention Study Dortmund- Continued (Coco)
Acronym: Coco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Child Nutrition, Dortmund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: RIChildNutrition
Record Dates: First submitted 2014-12-15; First posted 2015-01-22 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2015-05

CONDITIONS: Cognitive Function
Keywords: Having Lunch; Skipping Lunch

ARMS (2):
- having lunch/skipping lunch (Experimental): Lunch ad libitum on test day 1 and no lunch on test day 2. Water at libitum was constantly available on both days.
  Interventions: Other: Having lunch/skipping lunch
- skipping lunch/having lunch (Experimental): no lunch on test day 1 and lunch ad libitum on test day 2. Water at libitum was constantly available on both days.
  Interventions: Other: Skipping lunch/having lunch

INTERVENTIONS:
Other: Having lunch/skipping lunch — Lunch ad libitum on test day 1 and no lunch on test day 2. Water at libitum was constantly available on both days.
  Arms: having lunch/skipping lunch
Other: Skipping lunch/having lunch — No lunch on test day 1 and lunch ad libitum on test day 2. Water at libitum was constantly available on both days.
  Arms: skipping lunch/having lunch

SUMMARY:
The Cognition Intervention Study Dortmund (CogniDo) and the Cognition Intervention Study Dortmund PLUS (CogniDo PLUS) investigated the short-term effects of having school lunch versus skipping it on children's basal (CogniDo) and executive (CogniDo PLUS) cognitive functions in the afternoon. The present Coco study connect this two previous studies and investigates the effect of having school lunch versus skipping it on children's basal and executive cognitive functions later in the afternoon.

DETAILED DESCRIPTION:
Because of cerebral particularities, children may react highly sensitive to variations of nutrient supply. Therefore, an optimised composition of meals at favourable mealtime should be considered for optimal cognitive performance. The increasing implementation of all-day schools in Germany requires the children's catering for lunch at school. However, the number of 'meal skippers' is increasing among children and adolescents. Thus, the effect of skipping lunch at school on cognitive functioning is examined in this experimental cross-over trial. As prior intake of food can have an influence on the physiological effect of test meal, the children's dietary intake in the mid-morning is standardized. The intervention is integrated in everyday school life:

9.15 a.m. standardized snack within the frame of the regular break, 9.45 a.m. to 12.25 p.m. everyday school life, 12.25 p.m. either lunch (control) or water as a beverage (intervention of 'skipping meal'), 12.45 p.m. to 1.15 p.m. regular lunch break, 1.15 p.m. to 14.10 p.m. regular school lesson. 14.15 p.m. computerized tests of executive cognitive and basal (alertness) functioning, 3 p.m. lunch for the 'skipping meal'-group. Parameters of cognition with relevance to everyday school life are measured by a computerized test program developed by the Institute of Working Learning and Aging (ALA). Usual eating behaviour, sleep behaviour, physical activity and parental education were determined as control variables by questionnaires for children, parents.

ELIGIBILITY:
Inclusion Criteria:

* All fifth and sixth grade students of Gesamtschule Berger Feld with the consent of parents and child

Exclusion Criteria:

* Metabolic diseases or special diet

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Shifting: Change of total reaction time for a) [ms] | Participants were tested twice with one week wash out (1h after having/skipping lunch)
  Measuring global task-switching costs by a three-part computer trial.
  1. Non-switch: digits from 1 to 26 in random order are to put in order.
  2. Non-switch: Same as a) with letters from A to Z
  3. switch: digits 1 to 13 and letters A to M in random order to put in altering ascending order (digit, letter)
Shifting: Change of total reaction time for b) [ms] | Participants were tested twice with one week wash out (1h after having/skipping lunch)
  Measuring global task-switching costs by a three-part computer trial.
  1. Non-switch: digits from 1 to 26 in random order are to put in order.
  2. Non-switch: Same as a) with letters from A to Z
  3. switch: digits 1 to 13 and letters A to M in random order to put in altering ascending order (digit, letter)
Shifting: Change of total switch-costs [ms] | Participants were tested twice with one week wash out (1h after having/skipping lunch)
  Measuring global task-switching costs by a three-part computer trial.
  1. Non-switch: digits from 1 to 26 in random order are to put in order.
  2. Non-switch: Same as a) with letters from A to Z
  3. switch: digits 1 to 13 and letters A to M in random order to put in altering ascending order (digit, letter)
updating: change of ratio of missing [%] | Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
  Continuous monitoring and quick addition or deletion of contents within the working memory A sequence of 106 items (pictures of fruit and vegetables) is shown to the participants. A reaction is required if the actual shown item was equal to the item shown in the second to last.
updating: change of ratio of false alarms [%] | Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
  Continuous monitoring and quick addition or deletion of contents within the working memory A sequence of 106 items (pictures of fruit and vegetables) is shown to the participants. A reaction is required if the actual shown item was equal to the item shown in the second to last.
updating: change of mean reaction time [ms] | Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
  Continuous monitoring and quick addition or deletion of contents within the working memory A sequence of 106 items (pictures of fruit and vegetables) is shown to the participants. A reaction is required if the actual shown item was equal to the item shown in the second to last.
tonic alertness: change of mean reaction time [ms] | Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
  measures the level of alertness in response to a simple visual stimulus. Mean reaction time and the deviation of reaction time; subsidiary outcomes are the numbers of omission and commission errors.
tonic alertness: change of deviation of reaction time [ms] | Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
  measures the level of alertness in response to a simple visual stimulus. Mean reaction time and the deviation of reaction time; subsidiary outcomes are the numbers of omission and commission errors.
tonic alertness:change of numbers of omission and commission errors [n] | Time Frame: Participants were tested twice with one week wash out (1h after having/skipping lunch)
  measures the level of alertness in response to a simple visual stimulus. Mean reaction time and the deviation of reaction time; subsidiary outcomes are the numbers of omission and commission errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Child Nutrition, Dortmund, Dortmund, Germany